CLINICAL TRIAL: NCT01910454
Title: Cognitive Oriented Strategy Training Augmented Rehabilitation (COSTAR) Treatment Approach for Stroke
Acronym: COSTAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R03HD069626 (NIH)
Record Dates: First submitted 2013-07-22; First posted 2013-07-29 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: Stroke; Occupational Therapy; Cognition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Oriented Strategy Augmented Rehabilitation (COSTAR) (Experimental)
  Interventions: Behavioral: Cognitive-Oriented Strategy Augmented Rehabilitation (COSTAR)
- Task Specific Training (TST) (Active Comparator)
  Interventions: Behavioral: Task Specific Training (TST)

INTERVENTIONS:
Behavioral: Cognitive-Oriented Strategy Augmented Rehabilitation (COSTAR) — The protocol for COSTAR is based on the Cognitive-Orientation to daily Occupational Performance Intervention (CO-OP) approach which includes the following components: (1) Guided discovery - a process created by CO-OP to make certain that participants discover the strategies that will solve their own performance problems ; (2) Cognitive strategy use - participants are taught a global problem-solving strategy and are enabled to discover additional domain specific strategies that will support their skill acquisition and performance competence; and (3) Dynamic performance analysis - an observation-based process of identifying performance problems or performance breakdown. These three components from CO-OP are overlaid on the TST intervention protocol described above to address the overall hypothesis of this study: that an evidence-based stroke rehabilitation treatment protocol (task-specific training) can be enhanced when augmented with the catalyst of cognitive-oriented strategy use.
  Arms: Cognitive-Oriented Strategy Augmented Rehabilitation (COSTAR)
Behavioral: Task Specific Training (TST) — The protocol for task-specific training is based on criteria established by Winstein and Wolf (2008) who define task-specific training (TST) as a top-down approach to rehabilitation that is based on recent integrated models of motor control, motor learning, and behavioral neuroscience and that addresses skill acquisition of performance of meaningful and relevant tasks (Winstein and Wolf, 2008). Winstein and Wolf use current theory to identify three key ingredients for a task-specific training (pg 269): (1) Challenging enough to require new learning, and engagement with attention to solve the motor problem; (2) Progressive and optimally adapted such that over practice, the task-demand is optimally adapted to the patient's capability and the environmental context. The task should not be too simple or too repetitive nor too difficult; and (3) Interesting enough to invoke active participation through engagement in meaningful activity.
  Other Names: Task Oriented Training; Specific Task Training
  Arms: Task Specific Training (TST)

SUMMARY:
Stroke is the most serious disabling condition in the United States and the developed world. Novel stroke rehabilitation approaches, such as task-specific training, have shown promise in improving an individual's recovery in the rehabilitation setting; however, evidence suggests that these improvements are not generalized or transferred to the home, community, or work settings. Thus, these interventions usually do not impact overall health and participation outcomes. This research study seeks to improve task-specific training as a stroke rehabilitation approach by integrating it with evidence-based cognitive-oriented strategies which have shown great promise as a way to address the limitations of task-specific training. The new treatment protocol is called Cognitive-Oriented Strategy Training Augmented Rehabilitation, or COSTAR. The hypothesis of this study is that COSTAR will result in more efficient functional skill acquisition, better long-term retention of skills learned, and generalization and transfer of skills learned to home, community, and work settings.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older;
2. have completed all physician recommended rehabilitation and currently not receiving rehabilitation services;
3. at least one-month post-stroke;
4. have self-reported unmet functional goals; and
5. NIH Stroke Scale (NIHSS) total score of 2-12.

Exclusion Criteria:

1. have sustained a hemorrhagic stroke;
2. NIH Stroke Scale (NIHSS) aphasia rating of 1 or more (impaired speech);
3. MoCA cognitive screen score of less than 21 (impaired general cognitive ability);
4. neurological diagnoses other than stroke;
5. major psychiatric illness (bipolar disorder, OCD, panic disorder, PTSD, and/or borderline personality disorder);
6. no major depressive symptoms (PHQ-9 < 20);
7. a score of 6 or less on the CIHI aphasia screen combined items 64 and 66;
8. terminal illness;
9. blindness; and
10. non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Change from baseline to post-intervention (12 weeks)
Performance Quality Rating Scale (PQRS) | Change from baseline to post-intervention (12 weeks)

SECONDARY OUTCOMES:
Reintegration to Normal Living Index (RNLI) | Change from baseline to post-intervention (12 weeks)
Patient Reported Outcomes Measurement System (PROMIS-57) | Change from baseline to post-intervention (12 weeks)
Stroke Impact Scale (SIS) | Change from baseline to post-intervention (12 weeks)
Patient Health Questionnaire (PHQ-9) | Change from baseline to post-intervention (12 weeks)
Self-Efficacy Gauge (SEG) | Change from baseline to post-intervention (12 weeks)
Activity Card Sort (ACS) | Change from baseline to post-intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Wolf, OTD, MSCI, OTR/L, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis: Program in Occupational Therapy, St Louis, Missouri, United States

REFERENCES:
- [Background] Winstein, Carolee J, & Wolf, Steven L. (2009). Task-oriented training to promote upper extremity recovery. Stroke Recovery & Rehabilitation, 267-290.